CLINICAL TRIAL: NCT07308327
Title: Intestinal Probiotics Dietary Supplement
Brief Title: The Influence of Gut Microbiota on Ovarian Function: A Single-center, Randomized,Double Blind, Parallel-controlled, Exploratory Clinical Trial
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Songling Zhang (Other)
Responsible Party: Sponsor-Investigator, Songling Zhang, Doctor, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-HS-055
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Premature Ovarian Failure (POF)
Keywords: premature ovarian failure; intestinal bacteria
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, parallel-controlled, exploratory clinical trial was conducted on patients with ovarian dysfunction. The participants were randomly divided into two groups: Group A: received Akk. muciniphila bacteria, Group B: did not receive Akk. muciniphila bacteria. The clinical trial lasted for 3 months. Patients in Group A took one supplement of Akk. muciniphila bacteria daily. An early telephone visit was planned 15 days after supplementing with Akk. muciniphila bacteria (checking for abdominal distension, diarrhea, abdominal pain, nausea, vomiting, and changes in weight, etc.). Patients in Group B did not take Akk. muciniphila bacteria and were given a placebo (such as maltodextrin). The appearance and smell of the placebo were the same as the active bacterial supplement to avoid the introduction of bias through open-label. After 3 months, the samples were collected again at the hospital.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): health comparison
- POI/POF group (Experimental): Group A: Administered the Akk. muciniphila bacteria, Group B: Did not administer the Akk. muciniphila bacteria. A 3-month clinical trial was conducted.
  Interventions: Dietary Supplement: Akk Gut Bacteria Supplement; Other: Give a placebo

INTERVENTIONS:
Dietary Supplement: Akk Gut Bacteria Supplement — Taking the Aakk intestinal bacteria supplement for three months
  Arms: POI/POF group
Other: Give a placebo — The appearance and smell of the placebo are the same as those of the active bacterial agent.
  Arms: POI/POF group

SUMMARY:
In order to study the community profile of the intestinal microbiome in women with ovarian dysfunction, as well as the relationship between the changes in the intestinal microbiota and sex hormones, this study recruited 30 women with ovarian dysfunction and 30 healthy women. Sequencing was performed on the V3-V4 region of the 16S rDNA gene in fecal samples, and blood serum of the patients was collected for the study of changes in the systemic metabolome to reveal the significant differences in the intestinal microbiota between the subjects with ovarian dysfunction and the control group, as well as the related metabolic pathways.

DETAILED DESCRIPTION:
At the same time, in order to evaluate the effectiveness, safety and tolerance of supplementing the Akk. muciniphila bacteria, as well as to explore the impact of supplementing Akk. muciniphila bacteria on human ovarian function, this study aims to be the first clinical research to explore the effect of supplementing Akk. muciniphila bacteria on human ovarian function.

ELIGIBILITY:
Inclusion Criteria:

* 1. Ovarian dysfunction

  * Age < 40 years old; ② Irregular menstruation or amenorrhea for ≥ 4 months; ③ Two abnormal FSH levels (POF: FSH > 40 U/L; POI: FSH > 25 U/L); 2. Agree to participate in the study and be able to provide biological samples as required; 3. Body mass index within the normal range (18.5 kg/m² ≤ BMI < 24 kg/m²); 4. Strict contraception during treatment;

Control group:

1. Women have normal ovarian function;
2. No history of menstrual irregularity and infertility;
3. Regular menstruation;
4. Normal FSH levels (< 10 IU/L);
5. Age (< 40 years old) and body mass index (within the normal range 18.5 kg/m² ≤ BMI < 24 kg/m²) are matched with the case group; (The matching settings for the case group and the control group have been completed);

Exclusion Criteria:

* 1. Difficult to cooperate with researchers; 2. Those with congenital reproductive system disorders; 3. Those with chromosomal disorders; 4. Those with other systemic diseases; 5. Those with a history of ovarian surgery resection; 6. Chemotherapy/radiotherapy treatment; 7. Patients who have used antibiotics, antifungal drugs, antiviral drugs, proton pump inhibitors, corticosteroids or oral contraceptives within 3 months; 8. Patients who have been taking large doses of probiotic preparations for a long time.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
gonadal hormone concentrations | After taking the medicine for three months
Number of antral follicles | After taking the medicine for three months

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No